CLINICAL TRIAL: NCT02431039
Title: Comparison of Intraoperative Handling and Wound Healing Between NEOSORB Plus Antibacterial Suture With NEOSORB Suture: Prospective, Single-blind, Randomized Controlled Trial
Brief Title: Comparison Between NEOSORB Plus and NEOSORB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Medical Research Collaborating Center, Seoul, Korea (Other); Korea Health Industry Development Institute (Other Government); Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Principal Investigator, Chang Wook Jeong, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-1503-016-653
Record Dates: First submitted 2015-04-26; First posted 2015-04-30 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Skin Reaction to Suture Material

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEOSORB PLUS (Experimental): Subjects who are treated by NEOSORB PLUS
  Interventions: Device: NEOSORB PLUS
- NEOSORB (Active Comparator): Subjects who are treated by NEOSORB
  Interventions: Device: NEOSORB

INTERVENTIONS:
Device: NEOSORB PLUS — Fascia and subcutaneous tissue repaired by antibacterial suture materials (Chlorhexidine diacetate coated PGLA910)
  Other Names: Antibacterial suture material
  Arms: NEOSORB PLUS
Device: NEOSORB — Fascia and subcutaneous tissue repaired by non-antibacterial suture materials (PGLA910)
  Other Names: Non-antibacterial suture material
  Arms: NEOSORB

SUMMARY:
This study is to investigate whether NEOSORB Plus antibacterial suture (chlorhexidine diacetate coated PGLA910) is not inferior to NEOSORB suture (PGLA910) in the points of intraoperative handling.

DETAILED DESCRIPTION:
1. Enrollment

   1. Urologic surgery which needs fascia and subcutaneous tissue repairs
   2. Clean and clean-contaminated surgery
   3. Patients aged more than 18 years and under 80 years
2. Randomization

   1. NEOSORB Plus (chlorhexidine diacetate coated PGLA910) or NEOSORB (PGLA910) suture
   2. Stratification by operative methods: Open surgery vs. laparoscopic or robot-assisted laparoscopic surgery
3. Follow-up with 30 days

   1. Primary endpoint: intraoperative handling during operation
   2. Secondary endpoint: wound healing assessment on postoperative 1st (+1) days and 11th (± 4) days
   3. Safety evaluation: counting adverse events within postoperative 30 days

ELIGIBILITY:
Inclusion Criteria:

* Urologic surgery which needs fascia and subcutaneous tissue repairs
* Clean and clean-contaminated surgery

Exclusion Criteria:

* Contaminated surgery
* Wound requiring retention suture
* Suspicious malnutrition status
* Active infection status or AIDS
* Incision sites prone to expand, stretch, distend, or require support
* Allergy or hypersensitivity to chlorhexidine diacetate
* Significant active medical illness which in the opinion of the investigator would preclude protocol treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Overall handling | During the operation
  1 to 5 scale

SECONDARY OUTCOMES:
Ease of passage though tissue | During the operation
  1 to 5 scale
First-throw knot holding | During the operation
  1 to 5 scale
Knot tie-down smoothness | During the operation
  1 to 5 scale
Knot security | During the operation
  1 to 5 scale
Surgical hand | During the operation
  1 to 5 scale
Memory | During the operation
  1 to 5 scale
Lack of fraying | During the operation
  1 to 5 scale
Healing progress, apposition | On postoperative 1st(+1) and 11th(±4) day
  Complete vs. Incomplete
Infection | On postoperative 1st(+1) and 11th(±4) day
  No vs. YES
Seroma requiring drainage | On postoperative 1st(+1) and 11th(±4) day
  No vs. YES
Suture sinus, culture-negative | On postoperative 1st and 11(± 4)th day
  No vs. YES
Erythema | On postoperative 1st(+1) and 11th(±4) day
  0, + (closure line redness), ++(redness<2mm), +++ (redness>2mm)
Edema | On postoperative 1st(+1) and 11th(±4) day
  0, + (slight increase in firmness), ++(skin dimples with pressure), +++ (tense firmness)
Pain | On postoperative 1st(+1) and 11th(±4) day
  0, + (with pressure), ++(with touching), +++ (constant)
Skin temperative increase | On postoperative 1st(+1) and 11th(±4) day
  0, + (slight), ++(definite), +++ (hot, radiating)
30 days cumulative skin infection rate | Within postoperative 30 days
  No vs. YES
30 days cumulative seroma requiring drainage rate | Within postoperative 30 days
  No vs. YES
30 days cumulative suture sinus (culture-negative) rate | Within postoperative 30 days
  No vs. YES
Adverse events | Within postoperative 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Chang Wook Jeong, M.D.,Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Tae BS, Park JH, Kim JK, Ku JH, Kwak C, Kim HH, Jeong CW. Comparison of intraoperative handling and wound healing between (NEOSORB(R) plus) and coated polyglactin 910 suture (NEOSORB(R)): a prospective, single-blind, randomized controlled trial. BMC Surg. 2018 Jul 6;18(1):45. doi: 10.1186/s12893-018-0377-4. PMID 29980202